CLINICAL TRIAL: NCT05706753
Title: An Open-label, Non-randomized Study to Investigate the Effects of Twice-Daily Milvexian Administration on the Pharmacokinetics of Single Doses of Midazolam, Ethinylestradiol and Drospirenone in Healthy Adult Females
Brief Title: A Study of Milvexian in Healthy Adult Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Collaborators: Bristol Myers Squibb Company (BMS) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109284; 2022-002828-12 (EudraCT Number); 70033093THR1009 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy Female
MeSH Terms: interventions — milvexian; Midazolam; Ethinyl Estradiol; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Milvexian + Midazolam + Ethinylestradiol/Drospirenone (Experimental): Participants will receive midazolam on Day 1 and Day 19; ethinylestradiol and drospirenone on Day 2 and Day 20; and milvexian from Day 7 to Day 24.
  Interventions: Drug: Milvexian; Drug: Midazolam; Drug: Ethinylestradiol; Drug: Drospirenone

INTERVENTIONS:
Drug: Milvexian — Milvexian will be administered orally.
  Other Names: JNJ-70033093; BMS-986177
Drug: Midazolam — Midazolam will be administered orally.
Drug: Ethinylestradiol — Ethinylestradiol will be administered orally.
Drug: Drospirenone — Drospirenone will be administered orally.

SUMMARY:
The purpose of this study is to measure the effect of milvexian given for approximately 2 weeks on (a) how the liver metabolizes other drugs (in this case one called midazolam), and (b) the pharmacokinetics (the way the body absorbs, distributes, and gets rid of a drug) of an oral contraceptive pill in healthy adult females.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, and vital signs, and 12-lead electrocardiography (ECG) performed at screening and on 1 day prior midazolam intervention (Day -1)
* Healthy on the basis of clinical laboratory tests performed at screening and on Day -1 (screening) of the treatment phase. If the results of the serum chemistry panel, coagulation (activated partial thromboplastin time [aPTT] and prothrombin time [PT]), hematology, or urinalysis
* Body weight not less than 50.0 kilograms (kg) and body mass index (BMI; weight (kg) per height metered square (kg/m^2) within the range 18.5-30.0 kg/m^2 (inclusive) at screening and Day -1
* All women must have a negative highly sensitive serum human chorionic gonadotropin (beta-hCG) test at screening and urine pregnancy test on Day -1
* A woman must be: a. Not of childbearing potential or b. Of childbearing potential and practicing a highly effective method of contraception and agrees to remain on a highly effective method (failure rate of less than [<]1 percentage [%] per year when used consistently and correctly) until 4 days (5 half-lives) after last dose of milvexian-the end of relevant exposure

Exclusion Criteria:

* History of any known illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study intervention to the participant or that could prevent, limit or confound the protocol specified assessments
* History of any clinically significant drug or food allergies (such as anaphylaxis or hepatotoxicity) and known allergy to the study intervention or any of the excipients of milvexian, midazolam, or Drospifem 20 (ethinylestradiol + drospirenone)
* Clinically significant abnormal values for hematology, coagulation, clinical chemistry or urinalysis at screening or on Day -1 as determined by the investigator or appropriate designee. If any of the following laboratory rules are met at screening or Day -1, the participant should be excluded. A retest is allowed once: hemoglobin or hematocrit < lower limit of normal, platelet count < lower limit of normal, aPTT or PT greater than (>) 1.2 x upper limit of normal (ULN)
* Received an investigational intervention or used an invasive investigational medical device within 60 days or received a biological product within 3 months, or within a period less than 6 times the drug's half-life, if known, whichever is longer, before the first dose of study intervention or is currently enrolled in an investigational study
* Has used hormonal contraception injections or implants within 6 months of the first study intervention administration or has used any other hormonal contraception within 30 days of the first study intervention administration on Day 1

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Midazolam and 1-hydroxymidzolam | Up to Day 19
  Cmax is defined as the maximum observed plasma concentration of midazolam and 1-hydroxymidzolam.
Area Under the Plasma Concentration-time Curve from Time 0 to Time of the Last Observed Quantifiable Concentration (AUC[0-last]) of Midazolam and 1-hydroxymidzolam | Up to Day 19
  AUC(0-last) is defined as area under the plasma concentration-time curve from time 0 to time of the last observed quantifiable concentration of midazolam and 1-hydroxymidzolam.
Area Under the Plasma Concentration-time Curve from Time 0 to Infinite time (AUC[0-infinity]) of Midazolam and 1-hydroxymidzolam | Up to Day 19
  AUC(0-infinity) is defined as the area under the plasma concentration-time curve from time 0 to infinite time of midazolam and 1-hydroxymidzolam.
Maximum Observed Plasma Concentration (Cmax) of Ethinylestradiol and Drospirenone | Up to Day 25
  Cmax is defined as the maximum observed plasma concentration of ethinylestradiol and drospirenone.
Area Under the Plasma Concentration-time Curve from Time 0 to Time of the Last Observed Quantifiable Concentration (AUC[0-last]) of Ethinylestradiol and Drospirenone | Up to Day 25
  AUC(0-last) is defined as area under the plasma concentration-time curve from time 0 to time of the last observed quantifiable concentration of ethinylestradiol and drospirenone.
Area Under the Plasma Concentration-time Curve from Time 0 to Infinite Time (AUC[0-infinity]) of Ethinylestradiol and Drospirenone | Up to Day 25
  AUC(0-infinity) is defined as the area under the plasma concentration-time curve of from time 0 to infinite time ethinylestradiol and drospirenone.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Milvexian | Up to Day 19
  Cmax is defined as the maximum observed plasma concentration of milvexian.
Maximum Observed Plasma Concentration of Milvexian at Steady-state (Cmax,ss) | Up to Day 19
  Cmax,ss is defined as the maximum observed plasma concentration of milvexian at steady-state.
Area Under the Plasma Concentration-time Curve from Time 0 to Time of the Last Observed Quantifiable Concentration (AUC[0-last]) of Milvexian | Up to Day 19
  AUC(0-last) is defined as area under the plasma concentration-time curve from time 0 to time of the last observed quantifiable concentration of milvexian.
Area Under the Plasma Concentration-time Curve of Milvexian over the Dosing Interval (tau) at Steady-state (AUCtau,ss) | Up to Day 19
  AUCtau,ss is defined as the area under the plasma concentration-time curve of milvexian over the dosing interval (tau) at steady-state (AUCtau,ss).
Number of Participants with Adverse Events (AEs) | Up to 16 weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Number of Participants with Adverse Events (AEs) of Interest | Up to 16 weeks
  AEs of Interest includes bleeding events, liver enzyme elevation and clinical liver events, and cutaneous events.
Number of Participants with Abnormalities in Vital Signs | Up to 16 weeks
  Number of participants with abnormalities in vital signs (including blood pressure, pulse/heart rate, respiratory rate, body temperature) will be reported.
Number of Participants with Abnormalities in Electrocardiograms (ECGs) | Up to 16 weeks
  Number of participants with abnormalities in ECGs will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 16 weeks
  Number of participants with abnormalities in clinical laboratory tests will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium ClinicalTrial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- SGS Belgium NV, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency